CLINICAL TRIAL: NCT00679744
Title: A Dose-Escalated, Double-Blind, Placebo-Controlled, Randomized Phase I Clinical Trial of Pyrimethamine in Patients Affected With Chronic GM2 Gangliosidosis (Tay-Sachs or Sandhoff Variants)
Brief Title: A Phase I Study of Pyrimethamine in Patients With GM2 Gangliosidosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of funding
Sponsor: Exsar Corporation (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other); NYU Langone Health (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: 3448; CL-Pyrimethamine-001; FDA OPD Grant: FD-R-03448-01
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: G(M2) Ganglioside; Tay-Sachs Disease Ganglioside; Sandhoff Disease Ganglioside
Keywords: Tay-Sachs disease.; Sandhoff disease.; GM2 Gangliosidosis.; β-hexosaminidase deficiency.; Hexosaminidase; Phase I clinical trial.
MeSH Terms: conditions — Tay-Sachs Disease; Sandhoff Disease; Gangliosidoses, GM2 | interventions — Pyrimethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4 dose levels (Active Comparator): Pyrimethamine at 6.25, 12.5, 25 and 37.5 mg/day will be evaluated sequentially, starting from 6.25 mg/day. Escalation from 6.25 mg/day to 12.5 mg/day, and from 12.5 mg/day to 25 mg/day, will not perform until all patients in the previous dose cohort have been treated for 4 weeks and until results obtained 4 weeks after treatment initiation do not reveal toxicity. Additionally, escalation from 25 mg/day to 37.5 mg/day will not perform until all patients in the 25-mg/day cohort have been treated for 8 weeks, and until results obtained 4 weeks after the 8-week treatment do not reveal toxicity. Dose escalation is considered complete, if 2 patients experience a Grade 3 Adverse Event (AE) or if 1 patient experiences a Grade 4 AE at a particular cohort.
  Interventions: Drug: Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine — Pyrimethamine will be given PO once daily for 8 consecutive weeks.

SUMMARY:
Adult Tay-Sachs disease and Sandhoff diseases are caused by deficiency of an enzyme called β-hexosaminidase A, or Hex A in short. This enzyme is located in a particular cellular component, called lysosomes, inside the brain cells. The reason that Hex A of patients with Adult Tay-Sachs disease or Sandhoff disease is deficient is because this enzyme had gone through mutation, resulting in it not working very well. In healthy people, Hex A efficiently breaks down GM2-ganglioside, which is a by-product from cells of our body. However, patients with Adult Tay-Sachs disease or Sandhoff disease cannot efficiently break down GM2-ganglioside in the body. Therefore, these patients have high levels of this by-product in the brain cells, which causes the brain to be unable to function normally.

There is a drug called Pyrimethamine. This drug is used by doctors to treat specific types of infections called malaria and toxoplasmosis. Our laboratory test tube studies have shown that Pyrimethamine can help the Hex A enzyme to function in a normal manner. If Hex A can function normally in presence of Pyrimethamine, this drug should be able restore the brain malfunction of these patients since Hex A can now efficiently break down GM2-ganglioside with Pyrimethamine treatment.

Although results from laboratory test tube studies are promising and Pyrimethamine should theoretically restore brain function of these patients, we do not know if Pyrimethamine is safe or if it would actually work in patients. This study is the first study (a Phase I study) of testing Pyrimethamine to treat Adult Tay-Sachs and Sandhoff diseases. The objective of this study is to see if Pyrimethamine is safe in these patients and to see if it can restore the brain function of these patients.

DETAILED DESCRIPTION:
Adult Tay-Sachs (TSD) and Sandhoff disease (SD) result from a deficiency of lysosomal heterodimeric β-hexosaminidase A (Hex A, αβ). These disorders are characterized by progressive neurological deterioration that mainly affects motor, cerebral and spinocerebellar function. They affect fewer than 1000 people in the United States. There is no effective treatment for these diseases.

Substantial evidence supports a disease model for TSD and SD which attributes pathology to decreased or absent Hex A levels in neuronal lysosomes of the brain. The problem in GM2 - gangliosidosis is the inability of the cell to metabolize GM2 gangliosides. When the residual activity of Hex A falls below a critical threshold level, GM2 ganglioside influx into the lysosome (the site of Hex A activity) exceeds the degradation rate and excess substrate continuously accumulates. Consequently, the lysosomes increase in size and number, giving rise to a storage disease.

The majority of the mutations in Hex A affect the ability of the enzyme to obtain and/or retain its native 3-dimensional fold in the endoplasmic reticulum (ER) where intracellular quality control is performed to retain and degrade defective enzymes. Pharmacological chaperones (PC)s are small molecules that can stabilize the native conformation of a mutant enzyme in the ER and allow it to escape the ER's quality control system and its associated degradation pathway (ERAD). PCs have the potential to act as drugs when they can stabilize the native conformation of a mutant enzyme.

In 2006 ExSAR applied for orphan drug designation from the FDA for Pyrimethamine (Pyrimethamine) for the treatment of patients affected with late-onset GM2-gangliosidosis. The application is pending the positive outcome of clinical trials. Pyrimethamine is an FDA-approved drug which readily passes the bloodbrain barrier (BBB). It is currently used to treat malaria and toxoplasmosis. Our in vitro cell-based studies with fibroblasts from these patients show that Pyrimethamine can function as a PC for Hex A and raise intracellular Hex A levels. Our hypothesis is that Pyrimethamine administered to adult TSD and SD patients can improve neurological function and health.

The over objective of the project is to assess the safety and tolerability of the drug. We first conduct a Phase I trial, which is the current study, using Pyrimethamine to treat patients affected with GM2-gangliosidosis. Hex A and B (αβ) activities in plasma and peripheral blood leukocytes will also be measured. The working hypotheses of the Phase I trial are that Pyrimethamine administered according to the regimen of the trial will be tolerated and safe and result in increased Hex A levels in blood and brain.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and genetically confirmed diagnosis of GM2 Gangliosidosis caused by β-hexosaminidase deficiency resulting from mutations in the HEX-A or HEX-B genes, which has been shown to respond to Pyrimethamine treatment in previous cell culture experiments (Maegawa et al. 2006).
* Must be 18 years of age or older to participate in the study.
* Able to understand and cooperate with the requirements of the study protocol.
* Mentally competent, have ability to understand and willingness to sign the informed consent form.
* Able to travel to the participating study site.
* Women of child-bearing potential must use accepted contraceptive methods, and must have a negative serum or urine pregnancy test within 2 days prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists.
* Laboratory values ≤2 weeks prior to randomization must be within acceptable range.
* Body weight >40 kg (88 pounds).

Exclusion Criteria:

* Serious medical illness, significant cardiac disease that would increase patients' risk for toxicity.
* Any hematologic or related abnormality, especially megaloblastic anemia, leukopenia, thrombocytopenia, pancytopenia, atrophic glossitis, hematuria, and disorders of cardiac rhythm, pulmonary eosinophilia, etc.
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Possible folate deficiency, such as individuals with malabsorption syndrome, alcoholism, or pregnancy, and those receiving therapy (such as phenytoin) affecting folate levels.
* Any complex disease that may confound treatment assessment.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because Pyrimethamine is a "Pregnancy Category C" product).
* Lactating females because of the potential for serious adverse reactions in nursing infants.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Unwilling or unable to follow protocol requirements.
* Known hypersensitivity reactions, intolerance or adverse reactions to Pyrimethamine or to the inactive ingredients (corn and potato starch, lactose, and magnesium stearate).
* Evidence of systemic infection, or anyone who in the opinion of the investigator would not be suitable for the study.
* Test positive for HIV.
* Test positive for hepatitis B or hepatitis C.
* Patients with a history of convulsive disorders, since these patients are very susceptible to the nervous system toxicity of Pyrimethamine.
* Patients receiving any other investigational treatment for any indication within the past 4 weeks prior to initiation of Pyrimethamine treatment.
* A history of cancer of any type, since Pyrimethamine may be carcinogenic.
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of Pyrimethamine treatment.
* Patients who are receiving antifolic drugs and drugs associated with myelosuppression, or patients who are receiving drugs, when used in combination with Pyrimethamine, have been reported to induce some degree of hepatotoxicity:
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is safety and tolerability, based on conventional laboratory and clinical assessments. | The primary outcome measure, which is safety and tolerability, will be assessed weekly during the 8-week treatment period and biweekly during the 4-week post-treatment period.

SECONDARY OUTCOMES:
The secondary outcome measure is to assess changes in β-hexosaminidase A and B activities in plasma and peripheral blood leukocytes. | The secondary outcome measure will be assessed weekly during the 4-week treatment period and at the end of the 4-week post-treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Almassian, Ph.D., Study Chair — Exsar Corporation
Locations (3):
- United States (2):
  - New York University, School of Medicine, Department of Neurology, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
- Division of Clinical & Metabolic Genetics, Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Maegawa GH, Tropak M, Buttner J, Stockley T, Kok F, Clarke JT, Mahuran DJ. Pyrimethamine as a potential pharmacological chaperone for late-onset forms of GM2 gangliosidosis. J Biol Chem. 2007 Mar 23;282(12):9150-61. doi: 10.1074/jbc.M609304200. Epub 2007 Jan 21. PMID 17237499